CLINICAL TRIAL: NCT00174278
Title: Treatment With Recombinant Human Growth Hormone (Genotonorm®) In Children With Short Stature Secondary To A Long Term Corticoid Therapy. A Study of Efficacy and Safety.
Brief Title: Treatment With Recombinant Human Growth Hormone Genotonorm (Registered) In Children With Short Stature Secondary
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 96-8123-018; A6281217
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Growth Hormone Deficiency; Growth Retardation
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

INTERVENTIONS:
Drug: Somatropin

SUMMARY:
To assess the effect of long-term treatment by Genotonorm on linear growth

ELIGIBILITY:
Inclusion Criteria:

* All the patients who have benefit during one year of a treatment by Genotonorm during the study 94-8123-014
* All patients who have stopped during one year will be included if a signed written informed consent

Exclusion Criteria:

* Endocrine disease, except well substituted hypothyroidism
* Other severe chronic diseases (e.g. diabetes mellitus, cardiac or liver insufficiency)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14
Dates: Start 1997-02; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The main efficacy variable is the height SDS (SEMPE) before and after treatment.
The standing height of the patients is measured during the inclusion visit and at each follow-up visit.
The height measurements are always performed at the same time of the day by
use of a wallmounted device (e.g. Harpenden Stadiometer).
Each child has to be measured three times, the mean of these measurements is recorded in the Case Report Form as the present height.
The body weight is measured by use of a balance scale.
Puberty stage is assessed (according to Tanner´s cotation) at the same visits as height is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Paris, France

REFERENCES:
- [Derived] David H, Aupiais C, Louveau B, Quartier P, Jacqz-Aigrain E, Carel JC, Simon D. Growth Outcomes After GH Therapy of Patients Given Long-Term Corticosteroids for Juvenile Idiopathic Arthritis. J Clin Endocrinol Metab. 2017 Dec 1;102(12):4578-4587. doi: 10.1210/jc.2017-01455. PMID 29029101
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=96-8123-018&StudyName=Treatment+With+Recombinant+Human+Growth+Hormone+Genotonorm+%28Registered%29+In+Children+With+Short+Stature+Secondary+